CLINICAL TRIAL: NCT07076355
Title: Evaluation of the Ultrasonography-Guidance for Botulinum Toxin Type A Injection Into Lateral Pterygoid Muscle in Patients With TMJ Anterior Disc Displacement With Reduction
Brief Title: Ultrasound-Guided Botulinum Toxin A Injection for TMJ Disc Displacement With Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rosie Abdulqahar Othman, Principal Investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-3-24-2126
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Anterior Disc Displacement
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-Guided Botulinum Toxin Type A Injection (Experimental): Patients in this arm received an ultrasound-guided injection of botulinum toxin type A (BTX-A) into the lateral pterygoid muscle to treat temporomandibular joint anterior disc displacement with reduction (ADDwR). The procedure was performed under local anesthesia with real-time ultrasonographic visualization to ensure accurate delivery and minimize complications.
  Interventions: Drug: Botulinum Toxin type a (Botox)

INTERVENTIONS:
Drug: Botulinum Toxin type a (Botox) — A single dose of 25 units of botulinum toxin type A (BTX-A) was injected into the lateral pterygoid muscle using ultrasonography-guided technique. The injection was performed under local anesthesia with patient monitoring.
  Other Names: BTX-A

SUMMARY:
This clinical trial was designed to evaluate the effectiveness of ultrasonography-guided botulinum toxin type A (BTX-A) injection into the lateral pterygoid muscle for the management of temporomandibular joint (TMJ) anterior disc displacement with reduction (ADDwR). Ten patients diagnosed with ADDwR participated in the study. Each patient received an ultrasound-guided injection of 25 units of BTX-A into the lateral pterygoid muscle under local anesthesia. Clinical evaluations were performed preoperatively and at 2, 6, 12, and 24 weeks postoperatively. Outcome measures included pain levels assessed by the Numerical Rating Scale (NRS), TMJ sounds (clicking) detected using a stethoscope, disc position assessed by MRI, mandibular function parameters such as lateral excursion and maximum interincisal opening, and the Fonseca's questionnaire scores. The results demonstrated a significant reduction in pain and TMJ sounds, improvement in disc position, and enhanced mandibular function over a 6-month follow-up period. These findings suggest that ultrasonography-guided BTX-A injection into the lateral pterygoid muscle is a safe and effective treatment option for patients with TMJ ADDwR.

DETAILED DESCRIPTION:
This study investigated the therapeutic potential of ultrasonography-guided botulinum toxin type A (BTX-A) injection into the lateral pterygoid muscle in patients diagnosed with temporomandibular joint (TMJ) anterior disc displacement with reduction (ADDwR). The intervention was performed under local anesthesia with patient monitoring. High-frequency ultrasonography was utilized to accurately identify the lateral pterygoid muscle and guide the injection to minimize risks to adjacent anatomical structures.

The study followed patients over a 6-month period to assess changes in TMJ-related pain, functional parameters, and disc position. Pain intensity was measured using the Numerical Pain Rating Scale (NPRS), joint sounds were assessed clinically and with a stethoscope, disc position was evaluated via MRI, and mandibular movements were assessed by measuring lateral excursion and maximum interincisal opening. Patient-reported outcomes were also evaluated using the Fonseca's questionnaire.

The findings demonstrated a significant reduction in TMJ pain and joint noises, as well as improved mandibular function and disc alignment during the follow-up period. No major complications were observed, supporting the safety and efficacy of ultrasound-guided BTX-A injections in managing ADDwR.

This research provides clinical evidence for a minimally invasive and precise technique to manage TMJ internal derangements and reduce the impact of hyperactive lateral pterygoid muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bilateral anterior disc displacement with reduction (ADDwR) using Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).
* Patients aged 18 years or older.
* Patients who did not respond to previous conservative treatments.

Exclusion Criteria:

* Known allergy to any components of botulinum toxin type A (BTX-A).
* Presence of temporomandibular joint (TMJ) hypermobility.
* History of TMJ surgery.
* Presence of any significant pathology around the TMJ.
* Pregnant women.
* Individuals with systemic diseases that may affect the TMJ or the procedure.
* Patients with blood coagulopathy.
* Patients with unilateral ADDwR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity on the Numerical Pain Rating Scale (NPRS) | Baseline (preoperative), 2 weeks, 6 weeks, 12 weeks, and 24 weeks post-injection
  The Numerical Pain Rating Scale (0-10) was used to assess changes in pain intensity from baseline to follow-up time frames, with higher scores indicating greater pain.

SECONDARY OUTCOMES:
Change in TMJ Clicking Sounds | Baseline and at 2, 6, 12, and 24 weeks.
  Joint sounds were assessed using a stethoscope and scored as absent, heard only with a stethoscope, or heard unaided. We also quantified the intensity of the clicking sound using a custom made digital stethoscope to measure the sound in decibel units.
Change in Maximum Interincisal Opening (MIO) | Baseline and at 2, 6, 12, and 24 weeks.
  Maximum interincisal opening (measured in millimeters) were recorded at each follow-up.
Change in Lateral Excursion of the Mandible | Baseline and at 2, 6, 12, and 24 weeks.
  Lateral excursion (measured in millimeters) was recorded on both sides.
Change in Disc Position on MRI | baseline (preintervention) and 12 weeks postintervention.
  Disc position was assessed using MRI and recorded as an angular measurement (degrees) relative to the condyle.
Change in Fonseca's Questionnaire Score | baseline (preintervention) and 24 weeks postintervention.
  Fonseca's questionnaire was used to evaluate TMJ dysfunction severity on a scale from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Rosie A Othman, Principal Investigator — Tanta University; Ibrahim M Nowair, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Ahmed G Abushahba, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Mohamed S Abdelghany Elbrol, Principal Investigator — Faculty of Medicine, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No